CLINICAL TRIAL: NCT05661513
Title: Inventory of the Management of Acute Community-acquired Pneumonia in the Pneumology Department of the Strasbourg University Hospitals
Brief Title: Inventory of the Management of Acute Community-acquired Pneumonia in Strasbourg University Hospitals
Acronym: PPAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8718
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2022-12

CONDITIONS: Infection, Lung Parenchyma
Keywords: Community-acquired Pneumonia; Infection, Lung parenchyma; Rhinovirus; Respiratory syncitial virus; Influenza virus; Streptococcus pneumoniae
MeSH Terms: conditions — Infections; Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute community-acquired pneumonia (CAP) refers to an acute infection of the lung parenchyma, occurring within the first 48 hours of hospitalization. It is a frequent, serious pathology with a strong economic impact. Viruses (rhinovirus, respiratory syncitial virus, influenza virus for the most common) and Streptococcus pneumoniae are the most frequently encountered pathogens. However, more than half of the PACs have no microbiological documentation. The management of CAPs is based on national and international recommendations. Several studies have shown imperfect compliance by clinicians with recommendations with a prognostic impact.

The various published studies insist on the variability of the incidence, the type of pathogen, the severity and the economic impact, depending on the series. They also insist on the need to know the local epidemiology, in particular microbiological, in order to adapt the recommendations.

DETAILED DESCRIPTION:
The objective of the study is to determine the epidemiological, clinical, biological and imaging characteristics of people admitted for acute community-acquired pneumonia.

ELIGIBILITY:
Inclusion criteria:

* Adult subject (≥ 18 years old),
* acute community-acquired pneumonia (< 48 hours after admission),
* admitted from the Emergency Department, consultation or home.
* Subject not objecting to the reuse of their data for scientific research purposes

Exclusion criteria:

* Expressed refusal to reuse data for scientific research purposes.
* bronchitis, acute nosocomial pneumopathy, secondary infection due to bronchial dilation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with acute community-acquired pneumonia (< 48 hours after admission),
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03-09 (Estimated)

PRIMARY OUTCOMES:
Retrospectively determine the epidemiological, clinical, biological and imaging characteristics of people admitted for acute community-acquired pneumonia | Files analysed retrospectively from January 01, 2015 to December 31, 2019 will be examined
  Retrospective analysis of health data from patients' medical records

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pneumologie - CHU de Strasbourg - France, Strasbourg, France